CLINICAL TRIAL: NCT03565978
Title: Evaluation of a Cardiac Care Solution for Post-Hospital Management in Primary and Secondary Care of Patients Diagnosed With Coronary Artery Disease
Brief Title: Cardiac Care Solution for Coronary Disease Follow up
Acronym: BAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Principal Investigator, Yong Huo, Director, Department of Cardiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAMA 0.1
Record Dates: First submitted 2016-04-03; First posted 2018-06-21 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: ST Segment Elevation Myocardial Infarction; Non-ST Segment Elevation Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAMA solution (Experimental): This group will use BAMA solution. This is an digital solution used for cardiac post-discharge management. It is an application installed on a tablet. This arm will use this application and also have usual outpatient follow up.
  Interventions: Device: BAMA solution
- Usual care (No Intervention): Not using the application installed on the tablet. Usual outpatient follow up.

INTERVENTIONS:
Device: BAMA solution — Use of BAMA cardiac post-discharge management solution for patients education and follow up management
  Arms: BAMA solution

SUMMARY:
This is a prospective, randomized controlled trial. The aim of the study is to evaluate the impacts of a cardiac post-discharge management solution in the secondary prevention of Coronary Artery Disease (CAD).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the impacts of a cardiac post-discharge management solution in the population of cardiovascular (CVD) patients who were discharged from the hospital. The objectives include two parts:

Objective 1: Assess the feasibilities of using the solution by means of questionnaire.

Objective 2: Evaluate the impacts of the solution in the secondary prevention of Coronary Artery Disease (CAD).

Primary outcome: Compliance of coronary disease secondary prevention at 12 months.

Secondary outcome: Compliance of coronary disease secondary prevention at 6 months. Self-management behavior evaluation at the 6 and 12 months. Medication compliance at 6 and 12 months assessed by self-reporting questionnaire. Control rates of risk factors at the 6 and 12 months (serum LDL-C, blood pressure, fasting serum glucose); quality of life at the 6 and 12 months (EQ-5D, Seattle angina questionnaire); MACE (Major Adverse Cardiac Event) within 12 months (death, nonfatal myocardial infarction, nonfatal stroke, hospitalization for cardiac reason, unplanned coronary revascularization).

The study will be a two arm, randomized control study. The intervention group will use an application installed on a Pad besides standard outpatient follow up, while the control group will receive standard outpatient follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with CAD, including either condition below: once diagnosed with myocardial infarction; or once accepted coronary artery interventional therapy;
* Participants willing to use self-management solution and complying with follow-up plan;
* At point of enrollment, the patients should be at least (>=18) years
* Basic reading skills (Chinese)

Exclusion Criteria:

* Participants that are enrolled in another interventional clinical trial
* Participants who refuse to sign informed consent or withdraw for specific reasons recorded
* Participants who have cognition disorder and unable to communicate normally
* Participants who cannot master basic mobile technology skills to operate a mobile application after training

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-04-08 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Compliance for coronary heart disease secondary prevention at 12 months | 12 months
  Proportion of patients who use standardized secondary prevention medication according to current guidelines.

SECONDARY OUTCOMES:
Medication compliance at the 6, 12 months using the MMAS-8 (The eight-item Morisky Medication Adherence Scale) | 6 and 12 months
  The Chinese version MMAS-8, a self-administered rating scale for assessing medication adherence, contains eight items. Each item is measuring a specific behavior and is not a determinant of adherence behavior. Response choices are yes/no for items 1-7 and a 5-point Likert response for the last item. Each response of "no" is rated as "1" and each "yes" is rated as "0" except for Item 5, in which each response of "yes" is rated as "1" and each "no" is rated as "0". For Item 8, responses "0", "1", "2", "3" and "4", are rated as "0", "0.25", "0.75", "0.75" and "1", respectively. The total score on the MMAS-8 can range from 0 to 8, where higher scores indicate higher adherence. The degree of adherence was determined according to the score resulting from the sum of all the correct answers: low adherence (<6 points), medium adherence (6 to <8 points), and high adherence (8 points). In this study, patients were considered adherent when they had a score equal to eight in the MMAS-8.
Control rates of risk factors at the 6, 12 months | 6 and 12 months
  Blood pressure, serum LDL-C level and fast serum glucose
Quality of life at the 6, 12 months (EQ-5D simple score) | 6 and 12 months
  The EQ-5D(EuroQol-5 Dimensions) is an established health-related quality of life instrument, used frequently in both clinical trials and health services research. The EQ-5D instrument classifies respondent's present-day health status in five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression); each dimension is represented by one question with three severity levels (no problems, some problems and severe problems). Scores for the five dimensions can be converted into a utility index score by applying the scores from preference weights elicited from the UK general population. This calculation produces a value between -0.59 and 1.00, and a value below 0 indicates a worse health condition than death. Higher scores indicate better health status.
Quality of life at the 6, 12 months (EQ-5D Visual Analog Score) | 6 and 12 months
  EQ-5D Visual Analog Score was used in the survey, with anchor points 0 (worst health state) and 100 (best health state). The scale consisted of a horizontal line where every 10th was marked and labelled 0, 10, 20,…, 100. The question was framed: "On the scale please point out which point best represents your own health state today."
Quality of life at the 6, 12 month (Seattle angina questionnaire) | 6 and 12 months
  The Seattle Angina Questionnaire (SAQ), a 19-item index, is a commonly used disease-specific instrument for assessing symptoms and their impact on daily life with CAD. SAQ comprises five domains: physical limitation (PL), anginal stability (AS), anginal frequency (AF), treatment satisfaction (TS), and the disease perception (DP). SAQ is scored by assigning each response an ordinary value, from 1 (the lowest level of functioning) to 10 (the highest level of functioning), and summing across items within each of the 5 dimensional scales. Scale scores are then transformed to a scale of 0 to 100 by subtracting the lowest possible scale score, dividing the remainder by the range of the scale, and multiplying that by 100. Higher scores on SAQ subscales indicate higher levels of functioning/satisfaction and fewer limitations. The Chinese version of SAQ has been shown to be a valid, responsive, and reliable instrument and has been used in clinical trials.
MACE within 12 months (death, nonfatal myocardial infarction, nonfatal stroke, hospitalization with heart problem, unexpected revascularization) | 12 months
  Record events and describe
Self-management behaviors evaluation at the 6, 12 months using a local questionnaire | 6 and 12 months
  The Coronary Heart Disease Self-Management Behavior Scale used the Likert 5-point scale method to investigate patients' self-management behavior over the past 3 months. This scale has been widely used in China for self-management behavior of patients with coronary heart disease. The measurement has a good reliability and validity. The scale has three dimensions: (1) The dimensions of daily management, including management of general life and bad habits; (2) The dimension of emotion management is the emotional cognition management; (3)The dimensions of medical management include management of symptom, first-aid, disease knowledge and treatment adherence. The scores of the items in each dimension add up and transform to represent the total score of the dimension; the sum of the dimension scores represents the total score of self-management behavior, which range from 0 to 100. The higher the score that patient had indicates the better self-management behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Division of Cardiology, Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Gong Y, Zheng B, Fan F, Yi T, Zheng Y, He P, Fang J, Jia J, Zhu Q, Jiang J, Huo Y. Effects on Adherence to a Mobile App-Based Self-management Digital Therapeutics Among Patients With Coronary Heart Disease: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Feb 15;10(2):e32251. doi: 10.2196/32251. PMID 34906924